CLINICAL TRIAL: NCT00978809
Title: Epley Maneuver vs. Semont Maneuver for Benign Paroxysmal Positional Vertigo (BPPV): Evaluating Treatment Effectiveness by Postural Stability - a Double Blinded Randomized Controlled Trial.
Brief Title: Effects of Physical Treatment on Postural Stability in Benign Paroxysmal Positional Vertigo (BPPV) Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: major difficulties recruiting patients
Sponsor: Assuta Hospital Systems (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Hellmann Ory, Maccabi Health Services
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BPPV-2; 2009051
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2011-06

CONDITIONS: Benign Paroxysmal Positional Vertigo
Keywords: BPPV; postural stability; Epley; Semont
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Semont (Active Comparator): BPPV patients treated by Semont maneuver by a physical therapist.
  Interventions: Other: Semont maneuver
- control (No Intervention): healthy volunteers.
- Epley maneuver (Active Comparator): BPPV patients treated with Epley maneuver by a physical therapist.
  Interventions: Other: Epley maneuver

INTERVENTIONS:
Other: Epley maneuver
  Other Names: canalith repositioning maneuver
  Arms: Epley maneuver
Other: Semont maneuver
  Other Names: liberatory manoeuvre
  Arms: Semont

SUMMARY:
The propose of this study is to compare two methods of physical treatment for benign paroxysmal positional vertigo, by evaluating treatment effects on postural stability.

The trail design is a double blinded randomized controlled trail, with each patient going through three evaluations: before treatment, 1 week after treatment and 60 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* medical referral for treating "vertigo"
* subject has short episodes of rotatory vertigo (up to 1 minute)
* subject has positive Hallpike-Dix test with typical nystagmus
* repeated Hallpike-dix test will show fatigability

Exclusion Criteria:

* Hallpike-Dix test produces vertigo without nystagmus
* subject has BPPV of the horizontal or anterior semi-circular canal
* subject has other known vestibular or neurologic condition
* subject has nystagmus of a different type
* subject has a cervical spine problem which prevents the utilization of Epley or Semont maneuvers
* subject is unable to stand for 1 minute
* subject gets pharmacologic treatment for vertigo while doing the postural stability evaluation
* subject is under 18 years old or a pregnant female or cannot obtain informed concent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
postural stability | 60 days post treatment

SECONDARY OUTCOMES:
subjective vertigo | 60 days post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Itshak Melzer, Dr, Study Chair — Ben-Gurion University of the Negev; Moshe Puterman, Dr, Study Director — Soroka University Medical Center
Locations (1):
- Maccabi health services, Beersheba, Israel

REFERENCES:
- [Background] Blatt PJ, Georgakakis GA, Herdman SJ, Clendaniel RA, Tusa RJ. The effect of the canalith repositioning maneuver on resolving postural instability in patients with benign paroxysmal positional vertigo. Am J Otol. 2000 May;21(3):356-63. doi: 10.1016/s0196-0709(00)80045-9. PMID 10821549
- [Background] Di Girolamo S, Paludetti G, Briglia G, Cosenza A, Santarelli R, Di Nardo W. Postural control in benign paroxysmal positional vertigo before and after recovery. Acta Otolaryngol. 1998 Jun;118(3):289-93. doi: 10.1080/00016489850183340. PMID 9655200